CLINICAL TRIAL: NCT06204861
Title: Effectiveness Study of Capacitive and Resistive Electric Transfer Therapy Combined With Balance Training on Chronic Ankle Instability
Brief Title: The Effect of Capacitive and Resistive Electric Transfer Therapy in Chronic Ankle Instability Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Sport University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023341H
Record Dates: First submitted 2024-01-03; First posted 2024-01-12 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2024-01

CONDITIONS: Chronic Ankle Instability; Capacitive and Resistive Electric Transfer Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Capacitive and Resistive Electric Transfer Therapy Group (Experimental): Participants underwent 30 minutes of treatment per session, three times per week for four weeks during the experiment.
  Interventions: Other: Capacitive and Resistive Electric Transfer Therapy
- Balance Training Group (Experimental): Participants underwent 30 minutes of training per session, three times per week for four weeks during the experiment.
  Interventions: Other: Balance Training
- Balance Training Combined with Capacitive and Resistive Electric Transfer Therapy Group (Experimental): Participants underwent 30 minutes of training and treatment per session, three times per week for four weeks during the experiment.
  Interventions: Other: Balance Training Combined with Capacitive and Resistive Electric Transfer Therapy

INTERVENTIONS:
Other: Capacitive and Resistive Electric Transfer Therapy — Participants received a 10-minute intervention in CAP mode followed by a 20-minute intervention in RES mode.
  Arms: Capacitive and Resistive Electric Transfer Therapy Group
Other: Balance Training — The training program consists of five exercises: single-limb stance, single-limb stance with ball toss, single-limb stance with kicking, step-down with a single-limb stance, and wobble board. The program is conducted three times a week, and the difficulty level is increased every two weeks. Before and following the training, a physiotherapist will lead a warm-up and stretching session.
  Arms: Balance Training Group
Other: Balance Training Combined with Capacitive and Resistive Electric Transfer Therapy — Participants received a 10-minute intervention in CAP mode followed by a 20-minute intervention in RES mode. However, the B+CRET group received balance training along with CRET treatment.
  Arms: Balance Training Combined with Capacitive and Resistive Electric Transfer Therapy Group

SUMMARY:
The goal of this clinical trial is to compare the applicability and effectiveness of capacitive and resistive Electric transfer (CRET) therapy in combination with balance training in improving ankle function, proprioception, and balance in patients with chronic ankle instability (CAI). The main questions it aims to answer are:

* Can CRET therapy expedite the rehabilitation process for patients with chronic ankle instability?
* Does the combination of CRET therapy and balance training yield superior efficacy to other interventions?

This study involved 31 physically active participants with unilateral ankle instability, comprising 19 males and 12 females. The participants were randomly assigned to one of three groups: the balance training group (B Group), the capacitive and resistive electric transfer group (CRET Group), and the balance training combined with the capacitive and resistive electric transfer group (B+CRET Group).

DETAILED DESCRIPTION:
B group received only the balance training program, CRET group received only the CRET therapy, and B+CRET group received both the balance training program and the CRET therapy. Each intervention group received 12 interventions, three times per week, for a total of four weeks. Participants were instructed not to participate in any other exercise or treatment program during the experiment. Measurements were taken by the same researcher before and after the intervention. All participants were fully informed of the experiment's purpose and procedures and provided voluntary informed consent to participate. 31 participants completed the experimental study three times per week for four weeks under the guidance of a physical therapist. Only data from individuals with a completion rate of 75% or higher were included in the analysis.

The technical line of this study was to collect basic information about the participants, including age, height, weight, injury history, etc., and perform Ankle Special Tests, One Leg Standing Test, modified Star Excursion Balance Test, and fill out the Ankle Joint Functional Assessment Tool. Then the intervention groups underwent 12 sessions. In both the CRET and B+CRET groups, participants received a 10-minute intervention in CAP mode followed by a 20-minute intervention in RES mode. However, the B+CRET group received balance training along with CRET treatment.

The data was processed and analysed using SPSS 29.0 and Excel before and after the experiment. For count data that conformed to a normal distribution, mean ± standard deviation was used to express them. One-way ANOVA was used to analyse pre- and post-intervention between-group differences, with two-way comparisons using Tukey's test. Paired-sample t-tests were used to analyse pre- and post-intervention within-group differences. The Kruskal-Wallis H test was used to analyse pre- and post-intervention between-group differences for data that did not conform to a normal distribution. Similarly, the Wilcoxon signed-rank test was used to analyse pre- and post-intervention within-group differences. A significant difference was indicated by P<0.05 for all statistical results.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years;
* At least 12 months between the initial sprain and the current experiment, the sprain occurred with symptoms of inflammatory reactions such as pain and swelling, resulting in the inability to engage in physical activity for at least 1 day, and the most recent ankle sprain was more than 3 months away from the experiment;
* The occurrence of a re-sprain or "sensory instability" condition after the initial sprain, as follows: a. "sensory instability": at least 2 times within 6 months from the experiment; b. re-sprain: 2 times or 2 times of the same ankle sprain " condition as follows: a. "Sensory destabilization": at least 2 times within 6 months from the experiment; b. Re-sprain: 2 or more sprains of the same ankle;
* Ankle Joint Functional Assessment Tool (AJFAT) score ≤ 26;
* No complaint of instability in the other ankle;
* No mechanical ankle instability, i.e., negative anterior drawer test and talar tilt test
* No intervention by any means of rehabilitation before participation in this experiment.

Exclusion Criteria:

* The presence of lower extremity fracture on either side;
* The presence of central or peripheral nervous system injury
* The presence of lower extremity surgery on either side.

Ages: 18 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-10-15 (Actual)

PRIMARY OUTCOMES:
Ankle Joint Functional Assessment Tool | Each subject was tested before the first intervention training and after the twelfth intervention training (4 weeks after the first intervention).
  The Ankle Joint Functional Assessment Tool (AJFAT) can accurately identify functional instability. It consists of a 12-item self-assessment of pain and swelling, the ability to walk on stairs and uneven surfaces, make sharp stops and changes in direction, muscle strength, and stability. Participants evaluated the affected lower limb in comparison to the healthy limb using a grading system with five levels (0-4 points each), resulting in a maximum score of 48 points. Scores of 26 or lower were considered indicative of functional ankle instability and were included in the study. The time, place, and testers of the test were kept consistent.
One Leg Standing Test | Each subject was tested before the first intervention training and after the twelfth intervention training (4 weeks after the first intervention).
  The participant stood with their affected foot closed and their contralateral knee flexed at 90°. A score of one was recorded if any of the following occurred: the participant's supporting foot shifted, the contralateral lower extremity touched the ground, or the body swung beyond the center. The patient's total score within half-minute was recorded. Three tests were performed, and the average value was calculated. Subjects removed their shoes and socks to eliminate tactile effects. The time, place, and testers of the test were kept consistent.
The modified Star Excursion Balance Test | Each subject was tested before the first intervention training and after the twelfth intervention training (4 weeks after the first intervention). The time, place, and testers of the test were kept consistent.
  The participant was instructed to extend the unsupported leg as far as possible in three directions while balancing on one leg. Before the test, the length of the lower limb was measured from the anterior superior iliac spine to the lower end of the medial tibial ankle using a vernier straightedge while the participant was lying flat. To prevent learning effects, each participant practiced each direction six times before the formal test. The evaluation index chosen was relative distance, which is calculated as the maximum distance extended in each direction divided by the length of the leg and multiplied by 100. The time, place, and testers of the test were kept consistent.

CONTACTS AND LOCATIONS:
Overall Officials: Lin Song, Principal Investigator — Beijing Sport University
Locations (1):
- Beijing Sport University, Beijing, Beijing Municipality, China